# CONSENT FORM OF RESEARCH PARTICIPANTS

# Sahiwal Teaching Hospital, Sahiwal

| Case no | Date: | Study center: |
|---|---|---|
| · · | us dexmedetomidine we | rative analgesic effectiveness of bupivacaine and ound infiltration in abdominal surgeries under |
| Name of Research supervisor: | | Dr. Muhammad Shahid |
| Designation: | | Associate Professor Anesthesia & ICU,<br>Sahiwal Teaching Hospital, Sahiwal. |
| Name of research in charge: | | Dr. Hafsa Tariq |
| Department: | | Anesthesiology Department, SAHIWAL Teaching Hospital, Sahiwal. |
| Contact No: 03 | 321-6935010 | |
| Purpose: | | |
| | | ffectiveness of bupivacaine and bupivacaine plus abdominal surgeries under General Anaesthesia. |
| Procedure: | | |
| Every patient consent for par | - | ourpose of the study and requested to give his/her |

#### Possible risks:

There is no harm to participants in this research project.

### **Possible Benefits:**

All the tests of the patients participated in this study will be guided for treatment.

#### **Financial Consideration:**

There will be no financial burden on the patient. The financial benefits gained will be free of cost testing for the participant.

## **Confidentiality:**

All the records will be confidential and identity will be treated with confidentiality. The result of the study will be published for scientific purpose.

## **Exit from study:**

Every participant will have all the rights of getting excluded from the study even if the consent form is signed.

#### **Authorization:**

| Ihave been informed | about the details and application of the study. I understand |
|---|---|
| completely. I understand t | hat the study will not involve me with hazards. I have gone |
| through the contents of the | Proforma and I am willing to cooperate for the completion of |
| this data. | |
| Name of Patient: | Name of Guardian: |
| Signature: | Signature: |
| | Research In-charge: |
| | Signature: |